CLINICAL TRIAL: NCT07389421
Title: School Meals in Denmark: Evaluation of a National School Meal Pilot Program on Children's Health, Learning and Well-being - a Natural Experiment
Brief Title: School Meals in Denmark
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: University of Southern Denmark (Other); The Novo Nordic Foundation (Other)
Responsible Party: Principal Investigator, Nikolai Nordsborg, Professor, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-25070631
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Childhood Obesity; Childhood Obesity Pevention; Well-being/Quality of Life; Diet Habits; Cognitive Abilities; Healthy
Keywords: physical health; well-being; learning; diet
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: This is a pragmatic, matched-pair, cluster-randomized study conducted as a natural experiment. Allocation to the school meal program is determined at the school and grade level by a national policy initiative and not by the investigators.
  Schools are matched in pairs based on socioeconomic and geographic characteristics. Within each matched pair, intervention effects are estimated by comparing classes at the same grade level across schools, where one school implements the school meal program and the matched school does not. Control classes are recruited pragmatically from the same schools at a different grade level than the intervention classes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control classes (Experimental): The classes will continue with their regular meals, e.g. lunch packages
  Interventions: Behavioral: School meal classes

INTERVENTIONS:
Behavioral: School meal classes — Natural experiment embedded within the Danish National School Meal Pilot Program (2025-2028), which offers free school meals to selected public schools.
  Children receive a free school-provided meal (typically lunch) five days per week. Meals vary across schools, as each school selects its own meal provider.
  All meals must comply with the Nordic Nutrition Recommendations and the Danish Food-Based Dietary Guidelines, with a focus on fish, whole grains, fruits and vegetables, access to drinking water, and the promotion of children's food literacy.

SUMMARY:
This study looks at how a national school meal program affects the health, well-being, and learning of Danish schoolchildren aged 10 to 15 years.

The study is part of the Danish National School Meal Pilot Program (2025-2028), which provides free school meals at selected public schools. Some school classes receive free school meals, while other classes do not and are used for comparison.

Children are followed for about 1.5 years. Information is collected before and after the program using simple health measurements, questionnaires about well-being, and age-appropriate cognitive tests.

The study also uses information from Danish national registers to better understand the children's background and to study longer-term outcomes related to health, education, and social conditions. In addition, the study examines whether school meal programs are cost-effective by comparing their costs with potential benefits for children and society.

The goal of the study is to find out whether free school meals can improve children's health, well-being, and learning, and help reduce social differences.

DETAILED DESCRIPTION:
School Meals in Denmark is a prospective, open-label, matched-pair cluster-randomized controlled study conducted as a natural experiment alongside the Danish National School Meal Pilot Program. As allocation to the national program is determined by the Danish Ministry of Children and Education and not by the investigators, the study evaluates the effects of school meals under real-world conditions without introducing an additional experimental intervention.

Approximately 3,200 children in grades 3, 4, and 7 from 32 public schools are included. Participating schools are matched in pairs based on socioeconomic and geographic characteristics using national statistical data. Recruitment includes schools implementing the program either at the middle grades or at the lower secondary level. At each school, intervention classes are identified at the grade level receiving school meals.

Control classes are recruited pragmatically from the same schools but at a different grade level than the intervention classes. Intervention effects are estimated by comparing classes at the same grade level across matched schools, where one school implements the school meal program at that grade and the matched school does not. This approach allows for within-school control recruitment while preserving between-school comparisons at the same grade level.

Data are collected at two time points over a follow-up period of approximately 1.5 years using a pre-post design. Outcomes include anthropometric measures (height, weight, body composition assessed by bioelectrical impedance), cardiovascular indicators (blood pressure and resting heart rate), tablet-based cognitive performance tests, and child-reported questionnaires on well-being and psychosocial functioning. Parents complete brief electronic questionnaires addressing their child's psychosocial functioning and dietary habits.

In addition, observations of school meal settings are conducted to assess food intake and food waste, and menu plans from meal providers are collected to evaluate nutritional quality and compliance with dietary guidelines.

The study is designed to generate robust evidence on the real-world effects of school meal programs on children's health, well-being, and learning outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All children attending 3rd, 4th or 7th grade in the recruited schools

Exclusion Criteria:

* No exclusion criteria will be applied

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3200 (Estimated)
Dates: Start 2026-02-11 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Well-being/health related quality of life | Baseline, 16-22 months
  Between group difference in change in the total summary score of health-related quality of life measured with the KIDSCREEN 27 child self-report questionnaire. Data is collected using an adapted video and speech assisted electronic version with a smiley scale for each answer. The questionnaire assesses the child's physical well-being (5 items), psychological well-being (7 items), peers and social support (4 items), and school environment (4 items). Autonomy and parent relation (7 items) are not used.

SECONDARY OUTCOMES:
Psychological functioning | Baseline, 16-22 months
  Between group difference in change in the total difficulties score of the Strengths and difficulties questionnaire. Assessed using child reported version of the Strengths and Difficulties Questionnaire. An overall total difficulties score is calculated, along with five subscale scores: emotional symptoms, conduct problems, hyperactivity/Inattention, relationship problems, and prosocial behavior.
Internalizing problems | Baseline, 16-22 months
  Between group difference in change in the internalizing problem score of the Strengths and difficulties questionnaire, calculated as the sum of the emotional symptoms and peer problems scales scores. Assessed using the child-reported version of the Strengths and Difficulties Questionnaire.
Externalizing problems | Baseline, 16-22 months
  Between group difference in change in the externalizing behavior score of the Strengths and difficulties questionnaire, calculated as the sum of conduct problems, hyperactivity/Inattention subscales scores. Assessed using the child-reported version of the Strengths and Difficulties Questionnaire.
Prosocial Behavior | Baseline, 16-22 months
  Between group difference in change in the prosocial behavior score of the Strengths and difficulties questionnaire. Assessed using the child-reported version of the Strengths and Difficulties Questionnaire.
Psychological functioning (2) | Baseline, 16-22 months
  Between group difference in change in the total difficulties score of the Strengths and difficulties questionnaire. Assessed using parent reported version of the Strengths and Difficulties Questionnaire. An overall total difficulties score is calculated, along with five subscale scores: emotional symptoms, conduct problems, hyperactivity/Inattention, relationship problems, and prosocial behavior.
Externalizing problems (2) | Baseline, 16-22 months
  Between group difference in change in the externalizing behavior score of the Strengths and difficulties questionnaire, calculated as the sum of conduct problems, hyperactivity/Inattention subscales scores. Assessed using the parent-reported version of the Strengths and Difficulties Questionnaire.
Internalizing problems (2) | Baseline, 16-22 months
  Between group difference in change in the internalizing problem score of the Strengths and difficulties questionnaire, calculated as the sum of the emotional symptoms and peer problems scales scores. Assessed using the parent-reported version of the Strengths and Difficulties Questionnaire.
Prosocial Behavior (2) | Baseline, 16-22 months
  Between group difference in change in the prosocial behavior score of the Strengths and difficulties questionnaire. Assessed using the parent-reported version of the Strengths and Difficulties Questionnaire.
WHO-5 Well-Being Index | Baseline, 16-22 months
  Between group difference in change in the 5-question self-report tool from the World Health Organization measuring subjective mental well-being over the past two weeks, assessing feelings like cheerfulness, calmness, and interest.
School environment | Baseline, 16-22 months
  Between group difference in change in the school environment (4 items) score of the KIDSCREEN 27 child self-report questionnaire. Data is collected using an adapted video and speech assisted electronic version with a smiley scale for each answer.
Peers and social support | Baseline, 16-22 months
  Between group difference in change in the peers and social support (4 items) score of the KIDSCREEN 27 child self-report questionnaire. Data is collected using an adapted video and speech assisted electronic version with a smiley scale for each answer.
Psychological well-being | Baseline, 16-22 months
  Between group difference in change in the psychological well-being (7 items) score of the KIDSCREEN 27 child self-report questionnaire. Data is collected using an adapted video and speech assisted electronic version with a smiley scale for each answer.
Physical well-being | Baseline, 16-22 months
  Between group difference in change in the physical well-being (5 items) score of the KIDSCREEN 27 child self-report questionnaire. Data is collected using an adapted video and speech assisted electronic version with a smiley scale for each answer.
Resting blood pressure in mmHg | Baseline, 16-22 months
  Between group difference in change in systolic and diastolic blood pressure.
Resting heart rate beats/min | Baseline, 16-22 months
  Between group difference in change in heart rate.
Fat mass in kg | Baseline, 16-22 months
  Between group difference in change in fat mass measured by a bioimpedance analysis (InBody 270).
Fat free mass in kg | Baseline, 16-22 months
  Between group difference in change in fat free mass measured by a bioimpedance analysis (InBody 270).
Fat mass index in kg/m2 | Baseline, 16-22 months
  Between group difference in change in fat mass index measured by a bioimpedance analysis (InBody 270).
Fat free mass index in kg/m2 | Baseline, 16-22 months
  Between group difference in change in fat free mass index measured by a bioimpedance analysis (InBody 270).
Fat-Free-Mass-to-Fat-Mass ratio | Baseline, 16-22 months
  Between group difference in change in FFM-to-FM ratio measured by a bioimpedance analysis (InBody 270).
% Fat Mass | Baseline, 16-22 months
  Between group difference in change in % FM in kg measured by a bioimpedance analysis (InBody 270).
Weight status in % | Baseline, 16-22 months
  Between group difference in change in prevalence of children with underweight, normalweight, overweight and obesity, based on the cutoffs defined by Cole et al. and the International Task Force of Obesity. Body weight is measured by a bioimpedance analysis (InBody 270) and height by using a portable stadiometer.
BMI z-score | Baseline, 16-22 months
  Between group difference in change in BMI z-score based on WHO references. Weight and height is measured using weight from the bioimpedance analysis (InBody 270) and a portable stadiometer, respectively.
Sustained attention | Baseline, 16-22 months
  Performance in neuropsychological assessment of sustained attention ability assessed as errors during a sustained test procedure (Cambridge Neuropsychological Test Automated Battery, Cambridge cognition, UK).
Spatial working memory | Baseline, 16-22 months
  Performance in neuropsychological assessment of spatial working memory assessed as errors and strategy during the test procedure (Cambridge Neuropsychological Test Automated Battery, Cambridge cognition, UK).
Inhibitory control | Baseline, 16-22 months
  Performance in neuropsychological assessment of inhibitory control assessed as errors during the test procedure (Cambridge Neuropsychological Test Automated Battery, Cambridge cognition, UK).
Cognitive flexibility | Baseline, 16-22 months
  Performance in neuropsychological assessment of cognitive flexibility assessed as errors during the test procedure (Cambridge Neuropsychological Test Automated Battery, Cambridge cognition, UK).
Fine motor control | Baseline, 16-22 months
  Performance in neuropsychological assessment of fine motor control assessed as endpoint accuracy during the test procedure (Cambridge Neuropsychological Test Automated Battery, Cambridge cognition, UK).
Processing speed | Baseline, 16-22 months
  Performance in neuropsychological assessment of processing speed as choice reaction time (Cambridge Neuropsychological Test Automated Battery, Cambridge cognition, UK).

CONTACTS AND LOCATIONS:
Overall Officials: Nikolai B Nordsborg, PhD, Principal Investigator — University of Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided
If yes: De-identified individual participant data (only collected data, never registry data) will be made available upon reasonable request, subject to approval by the data controllers and in accordance with Danish data protection legislation.